CLINICAL TRIAL: NCT06228027
Title: Prediction of the Mortality in Acute Calculous Cholecystitis. The ACME Project.
Brief Title: External Validation os the ACME Scoring System
Acronym: ACME_2
Status: Not yet recruiting | Type: Observational
Sponsor: Hospital del Mar (Other)
Responsible Party: Principal Investigator, Ana María González Castillo, Doctor, Hospital del Mar
Other Study IDs: External_ACME Validation
Record Dates: First submitted 2024-01-18; First posted 2024-01-29 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: Acute Cholecystitis
Keywords: Acute Cholecystitis; Cholecystectomy; Tokyo Guidelines; Postoperative Complications; Mortality; High-risk patient
MeSH Terms: conditions — Cholecystitis, Acute; Postoperative Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 90 Days
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Acute calculous cholecystitis (ACC) is the second most frequent surgical condition in emergency departments. The recommended treatment is surgical treatment (ST) and the accepted mortality is <1%, but in severe and/or fragile patients is higher. Despite the Tokyo Guidelines, there no consensus on who is the unfit patient for ST. A recent study has identified 4 risk factors that predicts the mortality in a 92% of patients (ACME) and could help to develop new guidelines in ACC. The aim of this study is to perfom an external validation of the new simplified scoring system for mortality in ACC.

DETAILED DESCRIPTION:
This is a prospective multicenter observational study of 10.000 adults with ACC during 2 consecutive years (2025/2026), including baseline demographic characteristics, comorbidity severity defined as Charlson Comorbidity Index (CCI), ASA Score, Tokyo Guidelines severity classification and the new ACME Scoring system. The primary outcome is to study the prediction of mortality of ACME score. Secondary outcomes include complications following Clavien-Dindo's classification, C-statistic, and ROC Curves.

ELIGIBILITY:
Inclusion Criteria:

* Acute Calculous Cholecystitis

Exclusion Criteria:

* Acute Cholangitis
* Chronic Cholecystitis
* Neoplasia
* Acute Pancreatitis
* Pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All the consecutive admisions with an acute calculous cholecystitis, independent on the treatment indicated, during 2025 and 2026.
Sampling Method: Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2025-01-01 (Estimated); Primary Completion 2027-01-01 (Estimated); Study Completion 2027-04-15 (Estimated)

PRIMARY OUTCOMES:
Mortality | Jan 2025- Dec 2026
  Describe the mortality in the cohort and its causes
Complications | Jan 2025- Dec 2026
  Describe the mortality in the cohort by Clavien-Dindo's classification
ACME's prediction of mortality | Jan 2025- Dec 2026
  To describe the prediction in a ROC Curve of ACME Scoring System with C-Statistic

CONTACTS AND LOCATIONS:
Overall Officials: Ana María González Castillo, PhD, Principal Investigator — Hospital del Mar

IPD SHARING:
Plan to Share IPD: No